CLINICAL TRIAL: NCT07236983
Title: Gut Microbiota (GM) Biodiversity in Patients With Solid Tumors Treated With Immune Checkpoint Inhibitors (ICIs): a Monocenter Prospective Study to Identify the Interactions Between GM and ICIs
Acronym: GM&ICI
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Angioletta Lasagna, Oncologist, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: GM&ICI
Record Dates: First submitted 2025-03-07; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor Cancer Treatment With Immunotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although it is a milestone in the treatment of solid neoplasms, Immunotherapy (ICI) is still burdened by low response rate to the treatment and the occurrence of immune-related adverse events (irAEs). Recently, many studies have suggested that the The diversity of the intestinal microbiota (GM) can modulate response to ICIs [1]. The GM would be able to produce several molecules that can influence the growth of cancer cells and modulate anti-cancer immunity.

Our project aims to investigate changes in the subject and its relationship to immunotherapy.

Dynamic changes in cytokines can be a indicator of increased or decreased toxin translocation bacterial and therefore of the greater or lesser integrity of the barrier intestinal. Define the influence of diet on changes in GM can also help us understand how to modify these factors to improve the outcome of the subject undergoing immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years
2. Life-expectancy ≥6 months;
3. All participants have signed the consent form before enrollment
4. Patients with cancer who have to start immunotherapy with or without chemotherapy/targeted therapy

Exclusion Criteria:

1. Patients reporting an intake of antibiotic therapy during the last 30 days (rifaximin therapy used in patients with hepatocellular carcinoma in order to decrease the occurrence of overt Hepatic Encephalopathy is permitted) or any probiotic therapy in the last 30 days
2. A personal history of autoimmune or inflammatory bowel disease
3. Any major intestinal surgery (including bariatric surgery) in the previous six months
4. Ongoing enteral or parenteral nutrition
5. Patients with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with solid tumors who have to start immunotherapy are eligible. All types of cancer and all types of immunotherapy (anti CTLA-4/anti-PD-1/anti-PD-L1/a combination of anti-CTLA-4 and anti-PD1) with or without chemotherapy or target therapies are included. The estimated sample size is 100 cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The difference in alfa and beta diversity of GM in the stool sample | After 3 weeks, after 12 weeks, after 24 weeks and in the case of progression disease

SECONDARY OUTCOMES:
The difference in alfa and beta diversity of GM in the stool sample | From time 0, baseline (at the start of ICIs) to the occurrence of irAEs
The difference in the cytokine profile in the blood sample | From time 0 baseline (at the start of ICIs) to the different time points (after 3 weeks, after 12 weeks, after 24 weeks and in the case of progression disease)
The predictive factors associated with response to treatment with ICIs will be measured related to QueMD questionnaire score for adherence to Mediterranean diet at baseline, difference in QueMD questionnaire score from baseline to week 12. | At the end of Cycle 3 or 4 (each cycle is 28 days)
  The predictive factors associated with response to treatment with ICIs will be measured related to QueMD questionnaire score for adherence to Mediterranean diet at baseline, difference in QueMD questionnaire score from baseline to week 12, baseline body composition assessed through CT scan images analysis skeletal muscle (SM), SM index (SMI) defined by height-normalized SM, visceral adipose tissue (VAT), VAT index (VATI) defined by height-normalized VAT, subcutaneous adipose tissue (SAT), VAT-SAT ratio (VAT/SAT), intramuscular adipose tissue (IMAT)], difference in body composition from baseline to week 12, baseline diagnosis of sarcopenia [defined by the presence of both reduced handgrip strength (below 27 Kg in men and 16 Kg in female) and reduced SMI (using validated sex- and BMI-specific cutoffs)] and baseline NRS-2002 score. Report BMI in kg/m^2
The predictive factors associated with development of irAEs will be measured related to QueMD questionnaire score at baseline, baseline body composition and sarcopenia diagnosis, and baseline NRS-2002 score | Baseline
  Baseline body composition assessed through CT scan images analysis skeletal muscle (SM), SM index (SMI) defined by height-normalized SM, visceral adipose tissue (VAT), VAT index (VATI) defined by height-normalized VAT, subcutaneous adipose tissue (SAT), VAT-SAT ratio (VAT/SAT), intramuscular adipose tissue (IMAT)], difference in body composition from baseline to week 12.
  Baseline diagnosis of sarcopenia [defined by the presence of both reduced handgrip strength (below 27 Kg in men and 16 Kg in female) and reduced SMI (using validated sex- and BMI-specific cutoffs)]. Report BMI in kg/m^2 IRAE is defined by the Common Terminology Criteria for Adverse Events, version 5.0. This grading system refers to the severity of the adverse event associatedwith cancer therapy as follows: grade 1, mild; grade 2, moderate; grade 3, severe; grade 4, life threatening; and grade 5, death
Difference in body composition from baseline to week 12, related to the difference in alfa and beta diversity of GM in the stool sample from baseline to week 12 | From baseline to week 12
  Baseline body composition assessed through CT scan images analysis skeletal muscle (SM), SM index (SMI) defined by height-normalized SM, visceral adipose tissue (VAT), VAT index (VATI) defined by height-normalized VAT, subcutaneous adipose tissue (SAT), VAT-SAT ratio (VAT/SAT), intramuscular adipose tissue (IMAT)], difference in body composition from baseline to week 12. Report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Oncologia, Pavia, Pavia, Italy